CLINICAL TRIAL: NCT03768583
Title: Effect of Sensory Motor Training With and Without Sports Shoes on the Dynamic Postural Control of Athletes With Chronic Ankle Instability
Brief Title: Analysis of Sensory Motor Training in Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sensory motor training
Record Dates: First submitted 2018-07-21; First posted 2018-12-07 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2018-07

CONDITIONS: Recruitment
Keywords: Postural Balace; Physioteraphy; Ankle Injuries; Electromyography
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group TSM ICT sneakers (Experimental): * ICT with sneaker
  * five weeks
  * twice a week
  * half hour.
  Interventions: Other: Group TSM ICT sneakers
- Group TSM ICT barefoot (Experimental): * ICT barefoot
  * five weeks
  * twice a week
  * half hour.
  Interventions: Other: Group TSM ICT barefoot
- Group TSM health barefoot (Experimental): * Health with sneaker
  * five weeks
  * twice a week
  * half hour.
  Interventions: Other: Group TSM health barefoot
- Group TSM health sneakers (Experimental): * Health barefoot
  * five weeks
  * twice a week
  * half hour.
  Interventions: Other: Group TSM health sneaker

INTERVENTIONS:
Other: Group TSM ICT sneakers — Sensory motor training with sneakers for volunteers with Chronic ankle instability, for five weeks, twice a week.
  Arms: Group TSM ICT sneakers
Other: Group TSM ICT barefoot — Sensory motor training without sneakers for volunteers with Chronic ankle instability, for five weeks, twice a week.
  Arms: Group TSM ICT barefoot
Other: Group TSM health sneaker — Sensory motor training with sneakers for volunteers with Chronic ankle instability, for five weeks, twice a week.
  Arms: Group TSM health sneakers
Other: Group TSM health barefoot — Sensory motor training without sneaker for volunteers with Chronic ankle instability, for five weeks, twice a week.
  Arms: Group TSM health barefoot

SUMMARY:
Introduction: Sensory motor training (STS) is part of rehabilitation and injury prevention in individuals with chronic ankle instability (ICS). The use of footwear during SST may interfere with neuromuscular responses, but little is known about the difference in motor control response when training is applied with the use of shoes or bare feet. Objectives: To establish the effect of sensory motor training with and without sports shoes on the dynamic postural control of athletes with chronic ankle instability. Materials and Methods: The study will be performed with athletes linked to the Athletics of the State University of Londrina, aged between 18 and 30 years, both sexes, with chronic ankle instability assessed using the Cumberland Ankle Instability Tool (CAIT) questionnaire. Dynamic postural control will be evaluated in Force Platform and muscle recruitment through the electromyography of the muscles: anterior tibial, lateral and medial gastrocnemius, long fibular, gluteus maximus and gluteus medius. After the evaluation the volunteers will be randomized into two groups: 1) barefoot sensory-motor training and 2) sensory motor training with sneakers. The two groups will develop the same protocol of sensory motor training consisting of exercises, for five weeks, twice a week. At the end of the training they will be re-evaluated and the data analyzed. Expected Results: It is expected to find better postural control in the group that will perform in barefoot sensory-motor training.

DETAILED DESCRIPTION:
The total sample was determined in 54 volunteers, distributed equally in two groups: Chronic Ankle Instability and Control. Each group will be randomized for sensory-motor training with sneakers and without sneakers.

Inclusion criteria: athletes of both sexes, aged between 18 and 30 years, with history of ankle sprain in the last 12 months, sensation of instability or "yielding" of the ankle and score determined by the CAIT <24 questionnaire, did not perform sensory-motor training or conventional physiotherapy in the last six months.

Exclusion criteria: presence of pain complaints at the time of evaluation, recurrence of sprain with acute inflammatory signs, painful complaints in the lower limbs, lower limb surgery with neurological, cardiovascular, rheumatologic, diabetes, altered plantar sensitivity.

Participants with chronic ankle instability and controls will be randomly assigned to the two treatment groups, through the program www.ramdom.com, in blocks in the two groups: Sensory Motor Training Group with Tennis (TSMT) and Group Training Sensory Motor Barefoot ( TSMD).

Scratchs:

Since this is a study with intervention in participants with chronic ankle instability, there is a risk of new sprain during sensorimotor training. In case it occurs, the participant will receive all the support of the team coordinated by the professor Christiane Guerino de Souza Macedo in the extension project: Physiotherapy from theory to practice.

Procedures:

Initially the participants will complete the demographic data sheet (age, weight, height, BMI, level of physical activity and dominance in the lower limbs) and history of lower limb injury. Will respond to the chronic ankle instability questionnaire CAIT-p. They will sign the informed consent form (TCLE).

Following, the Lunge test will be performed to analyze ankle mobility. The same will be developed with the participant in orthostatism in front of a wall, with a tape measure, the participant will begin the test with a distance of 2cm from the wall and will be incremented by 1cm each time until the greater distance is reached. You will perform maximum knee flexion without the heel lifting from the floor or assuming a valgus position, with the goal of bringing the knee up to the wall. The result will be established by means of the halux-wall distance.

Postural control and muscle recruitment of a lower limb with the same direction should not be assessed by force platform and electromyography, respectively. The evaluations are made for the blind and according to the order of the instruments and the use or not of the shoe.

The anchoring of electromyographic analysis electrodes is performed on the anterior tibialis muscle (TA), lateral gastrocnemius (GL), medial gastrocnemius (GM), long fibularis (FL), gluteus maximus (GMe) and gluteus maximus (GMa). There will be a screening of electrotherapy supplements and cleaning of the area with alcohol rubbing (Moraes et al., 2012). The electrodes will be attached to the previous muscular points, according to the guide.

After placement of the electrodes the participant will be positioned with the lower limb to be tested on one step (based on height of applied force platform) and perform a series of assactions per second for thirty seconds controlled by metronome. This evaluation will be done 3 times. With a rest period of one full day in each test.

For an evaluation of dynamic postural control (BIOMEC400, Sistema EMG do Brasil, SP Ltda.). On the platform will be placed the member with chronic instability of the ankle and perform squatting to 30 seconds. With a rest period of one morning between each sitting test. They will be carried out 3 times with sneakers and 3 times with bare feet.

At this moment, the main parameters of COP-based postural control are: The area of COP ellipse (A-COP in cm²) and the mean COP oscillation distance (VEL in cm / s) are the most indicated in the directions: anteroposterior (A / P) and medium-lateral (M / L). Results were calculated for an average of three trials.

ELIGIBILITY:
Inclusion criteria:

* athletes of both sexes
* aged between 18 and 30 years,
* with history of the first ankle sprain for at least 12 months,
* feeling of instability or "flaccidity" of the ankle
* score determined by the CAIT questionnaire of less than 24,
* have not undergone sensory-motor or conventional physiotherapy training in the last six months.

Exclusion Criteria:

* Withdrawal at the time of the evaluation,
* Recurrence of sprain accompanied by signs of inflammation, acute and painful complaints in the lower group,
* history of lower limb surgery, neurological, cardiovascular, rheumatologic, diabetes, altered plantar sensitivity.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Postural control response after intervention | twenty weeks
  Response of sensorial motor training in improving motor control in volunteers with chronic ankle instability or not. Will use force platform.

SECONDARY OUTCOMES:
Muscle recruitment response after intervention | twenty weeks
  Response of sensorial motor training in the muscular recruitment of volunteers with chronic ankle instability or not, and the difference in response when performed with sneakers or barefoot. Will use electromyography.
measurement ankle dorsiflexion | twenty weeks
  The dorsiflexion will be mensure with the Lunge test in centimeter

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Macedo, Principal Investigator — State University of Londrina
Locations (1):
- university hospital of the State University of Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hiller CE, Refshauge KM, Bundy AC, Herbert RD, Kilbreath SL. The Cumberland ankle instability tool: a report of validity and reliability testing. Arch Phys Med Rehabil. 2006 Sep;87(9):1235-41. doi: 10.1016/j.apmr.2006.05.022. PMID 16935061
- [Background] Konradsen L, Bech L, Ehrenbjerg M, Nickelsen T. Seven years follow-up after ankle inversion trauma. Scand J Med Sci Sports. 2002 Jun;12(3):129-35. doi: 10.1034/j.1600-0838.2002.02104.x. PMID 12135444
- [Background] Heleno LR, da Silva RA, Shigaki L, Araujo CG, Coelho Candido CR, Okazaki VH, Frisseli A, Macedo CS. Five-week sensory motor training program improves functional performance and postural control in young male soccer players - A blind randomized clinical trial. Phys Ther Sport. 2016 Nov;22:74-80. doi: 10.1016/j.ptsp.2016.05.004. Epub 2016 May 10. PMID 27620862